CLINICAL TRIAL: NCT05928767
Title: Evaluation of the Clinical Frailty Scale (CFS) as a Risk Factor of Mortality in Adult Patients ≤65 Years of Age Admitted to Intensive Care for Septic Shock.
Acronym: Woodstock
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Lens (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-02
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Frailty; Septic Shock
MeSH Terms: conditions — Frailty; Shock, Septic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to demonstrate that "frail" patients, defined as having a CFS score greater than or equal to 5, and "severely" frail patients, defined as having a CFS score between [6-7] as defined by Bagshaw et al (14), constitute an independent risk factor (RF) for mortality.

In the same way, as an exploratory study, we will try to find out whether clinical frailty constitutes a risk factor for extending the length of hospital stay, the risk of short/medium-term readmission, as has already been demonstrated for patients admitted to intensive care from all causes (15), or for impaired quality of life.

The objective is to have a better understanding of the implications and outcomes associated with pre-hospital frailty in young critically ill patients.

This analysis will also help to clarify prognoses and contribute to better decision-making on the intensity and proportionality of care, as well as providing better information and helping to manage the expectations of patients and their families in terms of survival prognosis and subsequent quality of life.

DETAILED DESCRIPTION:
Recent studies show the impact of frailty in a middle-aged or even young population of patients admitted to critical care in terms of mortality (13), and the persistent risk of impairment of physical and mental capacities after resuscitation (14). To date, few studies have looked at clinical frailty as a risk factor for mortality in a middle-aged or young population, more specifically those suffering from septic shock, which is already known to be a major factor in morbidity and mortality (15,16), with repercussions on long-term quality of life.

The aim of the study is to demonstrate that "frail" patients, defined as having a CFS score greater than or equal to 5, and "severely" frail patients, defined as having a CFS score between [6-7] as defined by Bagshaw et al (14), constitute an independent risk factor (RF) for mortality.

In the same way, as an exploratory study, we will try to find out whether clinical frailty constitutes a risk factor for extending the length of hospital stay, the risk of short/medium-term readmission, as has already been demonstrated for patients admitted to intensive care from all causes (15), or for impaired quality of life.

The objective is to have a better understanding of the implications and outcomes associated with pre-hospital frailty in young critically ill patients.

This analysis will also help to clarify prognoses and contribute to better decision-making on the intensity and proportionality of care, as well as providing better information and helping to manage the expectations of patients and their families in terms of survival prognosis and subsequent quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years and ≤ 65 years
* Patient admitted to intensive care - resuscitation
* Patient admitted for suspected or documented type 3 sepsis
* Presence of vasopressor amines to maintain MAP > 65mmHg despite filling
* Lactatemia ≥ 2 mmol/L on admission.

Exclusion Criteria:

* Patient moribund on admission
* Patients with severe pre-existing dementia and/or cognitive decline, suffering from severe neurodegenerative diseases that prevent the patient from living independently at baseline, including mental illness requiring institutionalisation, including acquired or congenital mental retardation, etc.
* Pregnant women or women in labour
* Patients under guardianship or curatorship
* Patients deprived of their liberty
* Patient and/or family unable to speak or understand French.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to intensive care will be studied for this study. Patients meeting the inclusion criteria and with no non-inclusion criteria will be included in the study after obtaining the patient's or relative's, if applicable, non-objection.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
To show that the frailty score on admission is a risk factor for mortality at D28, independent of known risk factors, in young patients admitted to intensive care (ICU) for sepsis or septic shock. | 28 days after inclusion
  The odds ratio of frail patients to non-frail patients for the risk of all-cause death at D28

SECONDARY OUTCOMES:
To study the association, independently of known risk factors, between the frailty score on admission and mortality at day 90. | 90 days after inclusion
  Time from admission to death or last news, censored at D90
To study the association, independently of known risk factors, between the frailty score on admission and length of hospital stay | 90 days after inclusion
  The time between admission to IS and live discharge from hospital, death is considered a concurrent risk, the data are censored at 90 days
To study the association, independently of known risk factors, between the frailty score on admission and the number of days with recourse to invasive therapies | 90 days after inclusion
  Number of days with mechanical ventilation, with amines, with recourse to extra-renal purification (EER) during the IS stay.
To study the association, independently of known risk factors, between the frailty score on admission and readmission to critical care or hospitalisation before D90, among patients discharged alive from ICU before D90. | 90 days after inclusion
  Readmission to critical care or hospitalisation before D90, among patients discharged alive from ICU before D90.
To study the association, independently of known risk factors, between the frailty score on admission and describe changes in frailty between ICU admission and D90 in patients alive at D90. | 90 days after inclusion
  Change in frailty score defined by the CFS (continuous) between admission and D90 (in hospital or at home).
To study the association, independently of known risk factors, between the frailty score on admission and describe quality of life at D90 in patients alive at D90. | 90 days after inclusion
  Quality of life measured by the EQ5D score at D90 (in hospital or at home).

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Ch Germon Et Gauthier, Béthune
  - CH Boulogne sur Mer, Boulogne-sur-Mer
  - CHU de Dijon, Dijon
  - CH de Lens, Lens
  - CHU Lille, Lille